CLINICAL TRIAL: NCT00000713
Title: A Phase I Clinical Trial To Evaluate the Toxicity, Antiviral and Immunomodulatory Effects of a Range of Doses of Ampligen in HIV-Infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 038; 11014 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Polyribonucleotides; HIV Seropositivity; Dose-Response Relationship, Drug; Drug Evaluation; Acquired Immunodeficiency Syndrome; ampligen; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; HIV Seropositivity; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — poly(I).poly(c12,U)

INTERVENTIONS:
Drug: Ampligen

SUMMARY:
To determine the safety of ampligen at several doses in HIV-infected patients who have not yet developed AIDS or advanced AIDS related complex (ARC). Biologic, antiviral, and immunologic effects will be studied.

Evidence indicates that a long period with no symptoms follows infection with HIV. Individuals who are infected with the virus could benefit from therapy with a drug that acts to kill the virus or to stimulate the immune system of the individual or both. The immune system is the means the human body has for fighting infections. Ampligen is a suitable drug for clinical trials against HIV because it has been shown to stimulate the immune system and to inhibit HIV in vitro (test tube) at drug levels that can be achieved without noticeable clinical side effects.

DETAILED DESCRIPTION:
Evidence indicates that a long period with no symptoms follows infection with HIV. Individuals who are infected with the virus could benefit from therapy with a drug that acts to kill the virus or to stimulate the immune system of the individual or both. The immune system is the means the human body has for fighting infections. Ampligen is a suitable drug for clinical trials against HIV because it has been shown to stimulate the immune system and to inhibit HIV in vitro (test tube) at drug levels that can be achieved without noticeable clinical side effects.

Individuals entered in the study are given ampligen by intravenous infusion once during the first week of the trial and twice a week during the following 8 weeks. The dose each individual receives is determined by the responses of earlier individuals. Each is followed for 12 weeks after the last dose of ampligen is given. Each individual maintains a daily diary listing any symptoms or problems that occur, such as headache, nausea, or change in appetite. Other anti-HIV drugs cannot be taken during the trial, and aspirin or acetaminophen should not be taken for more than 2 hours without consulting the research staff. Blood is drawn at intervals during the trial and follow-up and used to determine the effect of ampligen on the HIV and the immune system as well as to monitor any toxicity and side effects.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Short-course therapy (7 days) with oral acyclovir or ketoconazole.

Patients must have:

* Evidence of HIV infection as measured by a confirmed positive antibody test.
* A confirmed or pending HIV blood culture, and serum p24 antigen test.
* The ELISA test confirmed by a licensed Western blot analysis if they are asymptomatic.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Aspirin or acetaminophen beyond 72 hours without contacting investigator.
* Chemoprophylaxis for Pneumocystis carinii pneumonia (PCP).

Patients with the following are excluded:

* AIDS.
* AIDS related symptoms or with advanced ARC and < 200 CD4 cells/mm3 and at least two of the following:
* Weight loss in excess of 10 lbs or 10 percent of body weight within a 6-month interval.
* Temperature > 38.5 degrees C with or without night sweats, persisting for more than 14 consecutive days or more than 15 days in a 30-day interval.
* Diarrhea defined as = or > 3 liquid stools per day, persisting for more than 30 days without definable cause.
* Recurrent oral candidiasis as documented by morphology or by response to antifungal therapy.
* Patients cannot have active oral candidiasis at the time of entry into the study; they must be free of candidiasis from baseline 1 to enrollment.
* Multidermatomal herpes zoster within the past 2 years.
* Hairy leukoplakia within the past 3 years.

Prior Medication:

Excluded within 14 days of study entry:

* Other biologic response modifiers.
* Corticosteroids.
* Systemic antibiotics.
* Excluded within 30 days of study entry:
* Other antiretroviral agents.
* Excluded within 60 days of study entry:
* Ribavirin.
* Zidovudine.

Concurrent neoplasms other than basal cell carcinoma of the skin.

Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Study Completion 1992-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Ho, Study Chair
Locations (1):
- Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Armstrong JA, McMahon D, Huang XL, Pazin GJ, Gupta P, Rinaldo CR Jr, Schoenfeld DA, Gaccione P, Tripoli CA, Bensasi S, et al. A phase I study of ampligen in human immunodeficiency virus-infected subjects. J Infect Dis. 1992 Oct;166(4):717-22. doi: 10.1093/infdis/166.4.717. PMID 1527407